CLINICAL TRIAL: NCT03902561
Title: Risk Factors of Inadequate Bowel Cleansing in Inpatients: a Predictive Score
Brief Title: Risk Factors of Poor Bowel Cleansing in Inpatients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Other Study IDs: ANT-POL-2017-01
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Colon Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: one time colonoscopy in inpatients — All the inpatients with indication of colonoscopy will be prepared with 4 liters polyethylene glycol bowel cleansing prior to colonoscopy. Colonoscopy will be performed as regular practice under conscious sedation.
  Other Names: 4 liters of Polyethylene glycol bowel preparation

SUMMARY:
The main purpose of the study is to determine risk factors of poor bowel cleansing in inpatients after a split-dose high volume preparation with 4 liters of polyethylene glycol. The quality of colon cleansing will be measured by the Boston bowel cleansing scale (more than or equal to 2 points in each segment). The secondary aim is to design a predictive score of poor bowel cleansing.

DETAILED DESCRIPTION:
It is well-known that inpatient status is a risk factor of inadequate bowel preparation. However this is a very mixed group, coexisting multiple factors containing several risk factors, such as elderly, comorbidities, a variety of medications, physical inactivity… Predictive factors in this population are probably different to those identified in outpatients. There is no strong evidence about the influence of these factors on inpatient bowel cleansing.

The researchers will offer to participate in the study to inpatients scheduled for colonoscopy who meet all the inclusion criteria and none of the exclusion criteria. The researchers will explain the purpose of the study and will ask to sign the informed consent. They will give verbal and written information on the diet and the bowel cleansing solution to be taken. A questionnaire will be administered about predictors of inadequate bowel cleansing. Activity will be measured by using a pedometer and a physical performance test.

Patients will take a liquid diet the day before the examination and they will be prepared with 4 liters of polyethylene glycol in split-dose regimen: 2 liters the evening before the examination (at 19.00 hours) and 2 liters 5 hours before colonoscopy The bowel cleansing quality following Boston Bowel Preparation Scale will be assessed by the endoscopist during the colonoscopy.

The aim of this study is to figure out the risk factors of bowel cleansing of inadequate bowel preparation in inpatients.

The inclusion of a maximum of 10 variables in the multivariate analysis will be considered: age, sex, short test of physical performance, Charlson index, indication (urgent or scheduled), polymedication (≥ 5 drugs), exposure to tricyclic antidepressants, calcium antagonists or opioids, constipation (<3 deposits per week and one of the following defecatory efforts), number of steps. For a predetermined percentage of 25% of patients with inadequate preparation, the inclusion of 400 inpatients who undergo a colonoscopy will be required. If we estimate an inclusion of about 10 patients per week, an inclusion period of about 10 months would be required.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with an indication of a colonoscopy
* Age ≥ 18 years.

Exclusion Criteria:

* Patients with previous colon surgery
* Last colonoscopy with poor bowel preparation.
* Ileus, intestinal obstruction, megacolon.
* Poorly controlled hypertension (Systolic and diastolic blood pressure > 180 and > 100, respectively).
* Terminal renal failure (pre-dialysis or dialysis).
* Congestive heart failure (NYHA III-IV).
* Acute liver failure.
* Severe psychiatric illness.
* Pregnancy or breastfeeding.
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The researchers will offer to participate in the study to inpatients scheduled for colonoscopy who meet all the inclusion criteria and none of the exclusion criteria. The researchers will explain the purpose of the study and will ask to sign the informed consent. They will give verbal and written information on the diet and the bowel cleansing solution to be taken. A questionnaire will be administered about predictors of inadequate bowel cleansing. Activity will be measured by using a pedometer and a physical performance test.
  Patients will take a liquid diet the day before the examination and they will be prepared with 4 liters of polyethylene glycol in split-dose regimen: 2 liters the evening before the examination (at 19.00 hours) and 2 liters 5 hours before colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
The validated Boston Bowel Preparation Scale will be used to measure colon cleansing quality | 8 months
  The Boston Bowel Preparation Scale scores cleansing quality from 0 to 3 points per segment (distal colon, transverse colon and right colon). The maximum score is 9 and the lowest 0. A score equal or more than 2 points per segment is considered an adequate preparation for this segment.

SECONDARY OUTCOMES:
To design a predictive score of inadequate bowel preparation [Time Frame: 1 years][Designated as safety issue: No] | 8 months
  Variables independently associated with Bowel cleansing with be used to build a predictive score

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Z Gimeno Garcia, MD, PhD, Principal Investigator — Hospital Universitario de Canarias

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gimeno-Garcia AZ, Hernandez G, Aldea A, Nicolas-Perez D, Jimenez A, Carrillo M, Felipe V, Alarcon-Fernandez O, Hernandez-Guerra M, Romero R, Alonso I, Gonzalez Y, Adrian Z, Moreno M, Ramos L, Quintero E. Comparison of Two Intensive Bowel Cleansing Regimens in Patients With Previous Poor Bowel Preparation: A Randomized Controlled Study. Am J Gastroenterol. 2017 Jun;112(6):951-958. doi: 10.1038/ajg.2017.53. Epub 2017 Mar 14. PMID 28291237
- [Result] Gimeno-Garcia AZ, Baute JL, Hernandez G, Morales D, Gonzalez-Perez CD, Nicolas-Perez D, Alarcon-Fernandez O, Jimenez A, Hernandez-Guerra M, Romero R, Alonso I, Gonzalez Y, Adrian Z, Carrillo M, Ramos L, Quintero E. Risk factors for inadequate bowel preparation: a validated predictive score. Endoscopy. 2017 Jun;49(6):536-543. doi: 10.1055/s-0043-101683. Epub 2017 Mar 10. PMID 28282690
- [Result] Rotondano G, Rispo A, Bottiglieri ME, De Luca L, Lamanda R, Orsini L, Bruzzese D, Galloro G; SIED Campania PISCoPO study group investigators; Romano M, Miranda A, Loguercio C, Esposito P, Nardone G, Compare D, Magno L, Ruggiero S, Imperatore N, De Palma GD, Gennarelli N, Cuomo R, Passananti V, Cirillo M, Cattaneo D, Bozzi RM, D'Angelo V, Marone P, Riccio E, De Nucci C, Monastra S, Caravelli G, Verde C, Di Giorgio P, Giannattasio F, Capece G, Taranto D, De Seta M, Spinosa G, De Stefano S, Familiari V, Cipolletta L, Bianco MA, Sansone S, Galasso G, De Colibus P, Romano M, Borgheresi P, Ricco G, Martorano M, Gravina AG, Marmo R, Rea M, Maurano A, Labianca O, Colantuoni E, Iuliano D, Trovato C, Fontana A, Pasquale L, Morante A, Perugini B, Scaglione G, Mauro B. Quality of bowel cleansing in hospitalized patients undergoing colonoscopy: A multicentre prospective regional study. Dig Liver Dis. 2015 Aug;47(8):669-74. doi: 10.1016/j.dld.2015.04.013. Epub 2015 Apr 25. PMID 26028360
- [Result] Yadlapati R, Johnston ER, Gregory DL, Ciolino JD, Cooper A, Keswani RN. Predictors of Inadequate Inpatient Colonoscopy Preparation and Its Association with Hospital Length of Stay and Costs. Dig Dis Sci. 2015 Nov;60(11):3482-90. doi: 10.1007/s10620-015-3761-2. Epub 2015 Jun 21. PMID 26093612